CLINICAL TRIAL: NCT05461885
Title: Value of Gym-based Exercise Training for Young Adults Receiving Antipsychotic Medication: A Pragmatic, Single-blinded, Multicenter Randomized Controlled Trial
Brief Title: Value of Gym-based Exercise Training for Young Adults Receiving Antipsychotic Medication: The Vega Trial
Acronym: Vega
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Bolette Rafn, Postdoc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vega Trial
Record Dates: First submitted 2022-06-29; First posted 2022-07-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Affective Disorder; Psychosis
MeSH Terms: conditions — Mood Disorders; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vega Exercise Community (Experimental): Participants will be offered one hour of tailored supervised, gym-based exercise training three times per week for a period of four months. In addition, participants are offered free-of-charge membership to the gym for six months and are invited to take part in training classes and use fitness equipment provided by the gym to regular members. The supervised program is tailored to meet the needs and requirements of this particular group of young adults and will include three weekly sessions of moderate-to-high intensity and mobility exercises.
  Interventions: Behavioral: Supervised exercise
- Usual care (No Intervention): Participants will receive treatment as usual and be informed of the official physical activity guidelines as part of the information on group allocation. Moreover, they will be advised to continue their daily living, as they normally would do, not guiding them to other interventions neither preventing them to do so. In addition, participants in the usual care group will be given a subsidized membership including access to the exercise classes for four months after the 12 months follow up.

INTERVENTIONS:
Behavioral: Supervised exercise — The exercise sessions start with warm-up exercises, followed by 10-20 minutes resistance training (Part A), 10-20 minutes High Intensity Functional Training (HIFT) (Part B) and cool down. Instructors are allowed to make local adjustments as the delivery of the intervention is considered pragmatic. The participants can either perform the exercise together as one group, in pairs or one-by-one depending on individual needs and requests.
  Arms: Vega Exercise Community

SUMMARY:
This is a multicentre, pragmatic, randomised controlled trial to estimate the effect of a 4-month gym-based exercise training program on 1) patient-rated personal recovery (primary outcome), 2) Health-related quality of life, behavioral and functional symptoms, and cardiometabolic risk factors (secondary outcomes) in young adults with psychotic disorders.

Four-hundred antipsychotic-treated young adults (between the age of 18 and 35), who are capable to undertake an exercise program (potentially with a friend or family member where possible) will be recruited from outpatient treatment units and mental health services. Participants will be randomised to treatment as usual or exercise at a 2:1 ratio in favor of exercise. Outcomes will be measured at baseline and at 4, 6 and 12 months after randomisation, by researchers masked to participant allocation.

DETAILED DESCRIPTION:
Background:

Antipsychotic medications are associated with development of metabolic side-effects. Patients with schizophrenia have a four-fold higher prevalence of metabolic syndrome, and a two-to-three-fold higher risk of cardiovascular diseases compared to the general population. These factors may contribute to the premature mortality of 15-20 years observed in people with schizophrenia. The increased morbidity and mortality in people with mental illness can be explained by several risk factors, including physical inactivity.

Evidence suggests that exercise can have beneficial effects on multiple cardiometabolic outcomes, and improve clinical symptoms, quality of life, global functioning, and reduce negative and depressive symptoms in people with schizophrenia. In general, greater effects are seen for higher doses of aerobic exercise and motivational theory-based interventions supervised by exercise professionals. However, because of strict inclusion criteria, the external validity of existing studies is limited, and effectiveness studies are urgently needed

Objectives:

The primary objective is to determine the effectiveness of participation in a four-month supervised, gym-based exercise program among people treated with antipsychotic medication compared to usual care on patient-rated recovery (primary outcome).

Secondary objectives are to examine if the gym-based exercise program compared to usual care improves the following:

1. Mental health
2. Health-related quality of life
3. Behavioral and functional symptoms
4. Metabolic health

As tertiary objectives, we will investigate if:

1. Prolongation of subsidized gym membership in addition to motivational text messages (extended support) will be superior to subsidized gym membership alone (minimal support), and to treatment as usual in relation to post-intervention adoption of physical activity.
2. The exercise program impacts the quality of life and physical and mental health of the participants' primary relative.
3. Participation in the gym-based program is associated with a reduction in the participants' use of mental health care services.
4. The exercise program is cost-effective.

Design:

This is a multi-center, pragmatic, randomized (1:2) superiority trial to compare a 4-month, supervised, gym-based exercise training program to usual care. The pragmatic nature of the trial entails that it is designed to evaluate the effectiveness of interventions in real-life routine practice conditions.

In order to explore different ways to support sustainment (i.e., post-intervention adherence/adoption of physical activity), and to guide strategies to facilitate adherence, we will do "a study within a trial" (SWAT). Hence participants randomized to the intervention at baseline, will be randomized (allocation ratio 1:1) after four months to minimal vs. extended support with regards to sustainment of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a psychotic disorder (F20-F29 Schizophrenia, schizotypal and delusional disorders) or an affective disorder (F30-F39 Mood [affective] disorders)
* able to read and speak Danish or English

Exclusion Criteria:

* advised from participating in exercise training by their treating doctor

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Personal recovery | Baseline to four months
  15-item Questionnaire about the Process of Recovery

SECONDARY OUTCOMES:
Personal recovery | Baseline to six months and 12 months
  15-item Questionnaire about the Process of Recovery
Mental health | Baseline to four months
  Mental Component Summary from the Short-Form 12 (SF-12) Health survey
Health-related quality of life | Baseline to four, six and 12 months
  Short-Form 12 (SF-12) Health survey
Affective symptoms | Baseline to four, six and 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional distress
Physical Activity | Baseline to four, six and 12 months
  International Physical Activity Questionnaire short form (IPAQ-SF)
Internalized Stigma | Baseline to four, six and 12 months
  Internalized Stigma of Mental Illness Inventory (ISMI-9) short form
Use of substance (alcohol, cannabis, drugs) | Baseline to four, six and 12 months
  Measured by self-developed items with responses for each substance: "never used", "use less than once a month", "regular use", "harmful use"
Sleep | Baseline to four, six and 12 months
  Brief Pittsburgh Sleep Quality Index (B-PSQI)
Positive and negative symptoms | Baseline to four, six and 12 months
  Colorado Symptom Index (MCSI)
Loneliness | Baseline to four, six and 12 months
  Measured by a single item on a Likert scale of 4 levels: "During the past 12 months, have you felt lonely?"
Abdominal circumference | Baseline to four, six and 12 months
  Measured with tape measure
Body weight | Baseline to four, six and 12 months
  Measured on a scale
Skeletal muscle mass | Baseline to four, six and 12 months
  Measured by bioimpedance
Total body fat | Baseline to four, six and 12 months
  Measured by bioimpedance
Cardiorespiratory fitness | Baseline to four, six and 12 months
  measured with the modified Ekblom-Bak submaximal cycle ergometer test
Blood pressure | Baseline to four, six and 12 months
  measured by a digital blood pressure monitor
Resting heart rate | Baseline to four, six and 12 months
  measured by a heart rate monitor
High density lipoproteins (HDL) | Baseline to four, six and 12 months
  Taken from routine blood tests (mmol/l)
Low density lipoproteins (LDL) | Baseline to four, six and 12 months
  Taken from routine blood tests (mmol/l)
Triglycerides | Baseline to four, six and 12 months
  Taken from routine blood tests (mmol/l)
Glycosylated haemoglobin (HbA1c) | Baseline to four, six and 12 months
  Taken from routine blood tests (mmol/l)
C-reactive protein (CRP) | Baseline to four, six and 12 months
  Taken from routine blood tests (mg/L)

OTHER OUTCOMES:
Use of the subsidized membership | four to six months
  To explore if prolongation of subsidized gym membership in addition to motivational text messages (extended support) is superior to subsidized gym membership alone (minimal support), and to treatment as usual in relation to post-intervention adoption of physical activity measured by use of the subsidized membership (intervention group only)
Extended vs. minimal support for physical activity | four to six months
  To explore if prolongation of subsidized gym membership in addition to motivational text messages (extended support) is superior to subsidized gym membership alone (minimal support), and to treatment as usual in relation to post-intervention adoption of physical activity measured by the IPAQ-SF (both groups).
Quality of life of primary relatives to participants | Baseline to four, six and 12 months
  To explore the impact of the Vega Exercise Community on the quality of life measured by SF-12 of the participants' primary relative
Sleep of primary relatives to participants | Baseline to four, six and 12 months
  To explore the impact of the Vega Exercise Community on sleep (measured by B-PSQI) of the participants' primary relative
Mental health of primary relatives to participants | Baseline to four, six and 12 months
  To explore the impact of the Vega Exercise Community on mental health (measured by PROMIS Emotional Distress-Depression - Short Form 4a) of the participants' primary relative
Physical activity of primary relatives to participants | Baseline to four, six and 12 months
  To explore the impact of the Vega Exercise Community on physical activity (measured by IPAQ-SF) of the participants' primary relative
Utilization of mental health care services | 24 months and 60 months
  To explore differences between groups of participants' long-term use of mental health care services, specifically number of inpatient and outpatient mental health contacts, including mental health emergency departments obtained from medical records
Cost of the Vega Exercise Community | Baseline to four, six and 12 months
  To explore the intervention cost i.e., education of instructors and delivery of exercise classes
Cost-effectiveness of the Vega Exercise Community | Baseline to four, six and 12 months
  To explore the cost-effectiveness by comparing the cost and health-related quality of life, which will be measured by the EuroQol-5 Domain (EQ-5D)

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Mental Health Centre Copenhagen, Copenhagen
  - Mental Health Centre Glostrup, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rafn BS, Andersen MF, Sorensen V, Bjerre ED, Baandrup L, Vernal DL, Mors O, Knop FK, Wolf RT, Tolver A, Firth J, Nohr N, Skou ST, Ebdrup BH, Midtgaard J. Value of gym-based group exercise versus usual care for young adults receiving antipsychotic medication: study protocol for the multicenter randomized controlled Vega trial. BMC Psychiatry. 2023 Aug 30;23(1):634. doi: 10.1186/s12888-023-05086-z. PMID 37648977

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05461885/SAP_000.pdf